CLINICAL TRIAL: NCT03058198
Title: The Research on 89Zr-ABT806 PET Imaging in High Grade Glioma and Its Correlation to EGFRvIII
Brief Title: The Research on 89Zr-ABT806 PET Imaging in High Grade Glioma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Dongxiao Zhuang, Professor, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 81672476
Record Dates: First submitted 2017-02-11; First posted 2017-02-20 (Actual); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Glioma
Keywords: Glioma; PET; EGFR vIII; Multimodal neuronavigation; Molecular pathology; PET-CT; Neuronavigation
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High Grade Glioma (Experimental): We plan to perform PET scanning on the patients with high grade gliomas after the injection of the second generation of EGFR tracer ,89Zr-ABT806（1-2mCi）, which can be specifically binded to EGFR vⅢ . After fusing the PET and MRI images, we precisely obtained the tissue from the"hot-spot" on the PET image through multimodal-neuronavigation-guided tumor biopsy. EGFRvⅢ status was detected by Sanger sequencing to analyze the correlation with the 89Zr-ABT806 PET image qualitatively and quantitatively. The final goal was to detect EGFR vⅢ by noninvasive molecular imaging procedure for the clinical outcome prediction and the selection of EGFR-targeted therapies.
  Interventions: Diagnostic Test: 89Zr-ABT806 PET

INTERVENTIONS:
Diagnostic Test: 89Zr-ABT806 PET — Patients will be given IV bolus injection of 89Zr-ABT806(1-2mCi). The first 89Zr-ABT806 PET scan will be performed about 72 to 120 hours after injection of tracer. The second 89Zr-ABT806 PET scan will be performed about 120 to 168 hours after injection of tracer. Semi-quantitative analysis was performed using the maximum standardized uptake value (SUVmax) and T/N ratio.

SUMMARY:
The epidermal growth factor receptor variant Ⅲ(EGFR vⅢ) is commonly detected in high-grade gliomas, which is also an important epitope in EGFR-targeted therapies and correlated to poor prognosis. However, detection of this mutant usually needs resected tumor samples. For biopsy samples, test results may not represent the EGFR vⅢ status of the whole tumor tissues because of the heterogeneity of tumor. It is also not applicable for patients who are not suitable for surgical procedure due to the tumor location or patients' general conditions. Because of the importance of the epidermal growth factor receptor (EGFR) signal pathway in oncogenesis, maintenance, and progression of high grade glioma, there has been an intense effort to develop noninvasive molecular imaging approach for the selection and monitoring of EGFR-targeted therapies.

Based on investigators' previous study, investigators plan to perform PET scanning on the participants with high grade gliomas after the injection of the second generation of EGFR tracer ,89Zr-ABT806, which can be specifically binded to EGFR vⅢ . After fusing the PET and MRI images, investigators precisely obtain the tissue from the"hot-spot" on the PET image through multimodal-neuronavigation-guided tumor biopsy. EGFRvⅢ status will be detected by molecular methods to analyze the correlation with the 89Zr-ABT806 PET image qualitatively and quantitatively. Investigators' final goal is to detect EGFR vⅢ by noninvasive molecular imaging procedure for the clinical outcome prediction and the selection of EGFR-targeted therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical manifestations and imaging examination (CT, MRI, et al) are in accordance with high grade glioma
2. No PET/CT scanning contraindications
3. No MRI scanning contraindications
4. Patients older than 18 years old
5. ECOG score between 0 to 2
6. Patients with sufficient bone marrow, kidney and liver function reserve.
7. All patients gave written informed consent.

Exclusion Criteria:

1. Patient who has received immune therapy, radiation therapy, chemotherapy, hormone drugs, biological products or other clinical trials within 14 days.
2. Patient who has received EGFR monoclonal antibody therapy within 4 weeks.
3. Patients who has not fully recovered form the past drug toxicity reaction (CTCAE in grade 2 or above).
4. Patient who has received major surgery within 7 days.
5. Patients with allergies to immunoglobulin.
6. Breastfeeding women.
7. pregnant women
8. Patients with severe clinical condition.
9. Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity of 89Zr-ABT806 PET | 4 years
  After fusing the 89Zr-ABT806 PET and MRI images, investigators precisely obtained the tissue from the"hot-spot" on the PET image through multimodal-neuronavigation-guided tumor biopsy. EGFRvⅢ status will be analyzed by molecular methods. The sensitivity and specificity of 89Zr-ABT806 PET will be measured with statistic methods.

SECONDARY OUTCOMES:
The overall survival time of participants | 4 years
  regular follow-up
The progression-free survival time of participants | 4 year
  regular follow-up
The correlation between EGFRvIII mutation and prognosis of participants | 4 year

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan hospital, Fudan university, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wong AJ, Ruppert JM, Bigner SH, Grzeschik CH, Humphrey PA, Bigner DS, Vogelstein B. Structural alterations of the epidermal growth factor receptor gene in human gliomas. Proc Natl Acad Sci U S A. 1992 Apr 1;89(7):2965-9. doi: 10.1073/pnas.89.7.2965. PMID 1557402
- [Background] Ekstrand AJ, James CD, Cavenee WK, Seliger B, Pettersson RF, Collins VP. Genes for epidermal growth factor receptor, transforming growth factor alpha, and epidermal growth factor and their expression in human gliomas in vivo. Cancer Res. 1991 Apr 15;51(8):2164-72. PMID 2009534
- [Background] Libermann TA, Razon N, Bartal AD, Yarden Y, Schlessinger J, Soreq H. Expression of epidermal growth factor receptors in human brain tumors. Cancer Res. 1984 Feb;44(2):753-60. PMID 6318976
- [Background] Sugawa N, Ekstrand AJ, James CD, Collins VP. Identical splicing of aberrant epidermal growth factor receptor transcripts from amplified rearranged genes in human glioblastomas. Proc Natl Acad Sci U S A. 1990 Nov;87(21):8602-6. doi: 10.1073/pnas.87.21.8602. PMID 2236070
- [Background] Yamazaki H, Fukui Y, Ueyama Y, Tamaoki N, Kawamoto T, Taniguchi S, Shibuya M. Amplification of the structurally and functionally altered epidermal growth factor receptor gene (c-erbB) in human brain tumors. Mol Cell Biol. 1988 Apr;8(4):1816-20. doi: 10.1128/mcb.8.4.1816-1820.1988. PMID 3380099
- [Background] Malden LT, Novak U, Kaye AH, Burgess AW. Selective amplification of the cytoplasmic domain of the epidermal growth factor receptor gene in glioblastoma multiforme. Cancer Res. 1988 May 15;48(10):2711-4. PMID 2834047
- [Background] Ekstrand AJ, Sugawa N, James CD, Collins VP. Amplified and rearranged epidermal growth factor receptor genes in human glioblastomas reveal deletions of sequences encoding portions of the N- and/or C-terminal tails. Proc Natl Acad Sci U S A. 1992 May 15;89(10):4309-13. doi: 10.1073/pnas.89.10.4309. PMID 1584765
- [Background] Nagane M, Coufal F, Lin H, Bogler O, Cavenee WK, Huang HJ. A common mutant epidermal growth factor receptor confers enhanced tumorigenicity on human glioblastoma cells by increasing proliferation and reducing apoptosis. Cancer Res. 1996 Nov 1;56(21):5079-86. PMID 8895767
- [Background] Batra SK, Castelino-Prabhu S, Wikstrand CJ, Zhu X, Humphrey PA, Friedman HS, Bigner DD. Epidermal growth factor ligand-independent, unregulated, cell-transforming potential of a naturally occurring human mutant EGFRvIII gene. Cell Growth Differ. 1995 Oct;6(10):1251-9. PMID 8845302
- [Background] Nishikawa R, Ji XD, Harmon RC, Lazar CS, Gill GN, Cavenee WK, Huang HJ. A mutant epidermal growth factor receptor common in human glioma confers enhanced tumorigenicity. Proc Natl Acad Sci U S A. 1994 Aug 2;91(16):7727-31. doi: 10.1073/pnas.91.16.7727. PMID 8052651
- [Background] Pedersen MW, Tkach V, Pedersen N, Berezin V, Poulsen HS. Expression of a naturally occurring constitutively active variant of the epidermal growth factor receptor in mouse fibroblasts increases motility. Int J Cancer. 2004 Feb 20;108(5):643-53. doi: 10.1002/ijc.11566. PMID 14696090
- [Background] Lammering G, Hewit TH, Holmes M, Valerie K, Hawkins W, Lin PS, Mikkelsen RB, Schmidt-Ullrich RK. Inhibition of the type III epidermal growth factor receptor variant mutant receptor by dominant-negative EGFR-CD533 enhances malignant glioma cell radiosensitivity. Clin Cancer Res. 2004 Oct 1;10(19):6732-43. doi: 10.1158/1078-0432.CCR-04-0393. PMID 15475464
- [Background] Lammering G, Valerie K, Lin PS, Hewit TH, Schmidt-Ullrich RK. Radiation-induced activation of a common variant of EGFR confers enhanced radioresistance. Radiother Oncol. 2004 Sep;72(3):267-73. doi: 10.1016/j.radonc.2004.07.004. PMID 15450724
- [Background] Feldkamp MM, Lala P, Lau N, Roncari L, Guha A. Expression of activated epidermal growth factor receptors, Ras-guanosine triphosphate, and mitogen-activated protein kinase in human glioblastoma multiforme specimens. Neurosurgery. 1999 Dec;45(6):1442-53. doi: 10.1097/00006123-199912000-00034. PMID 10598712
- [Background] Emrich JG, Brady LW, Quang TS, Class R, Miyamoto C, Black P, Rodeck U. Radioiodinated (I-125) monoclonal antibody 425 in the treatment of high grade glioma patients: ten-year synopsis of a novel treatment. Am J Clin Oncol. 2002 Dec;25(6):541-6. doi: 10.1097/00000421-200212000-00001. PMID 12477994
- [Background] Li G, Wong AJ. EGF receptor variant III as a target antigen for tumor immunotherapy. Expert Rev Vaccines. 2008 Sep;7(7):977-85. doi: 10.1586/14760584.7.7.977. PMID 18767947